CLINICAL TRIAL: NCT02537366
Title: Dexmedetomidine for Non-invasive Ventilation After Chest Trauma (VENDETTA)
Brief Title: Dexmedetomidine for Non-invasive Ventilation After Chest Trauma
Acronym: VENDETTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EssaiClinique-VENDETTA
Record Dates: First submitted 2015-08-21; First posted 2015-09-01 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Thoracic Injuries
MeSH Terms: conditions — Thoracic Injuries | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Sodium Chloride 0,9 % Continuous IV infusion begun one hour before NIV session at 0.07 ml/kg/h Adaptation to sedation status by changing infusion speed of 0.02 ml/kg/h every 30 minutes up to 0.14 ml/kg/h Sedation objective Richmond Agitation Sedation Scale -3 (moderate sedation) to 0 (alert and calm)
  Interventions: Drug: Placebo
- DEX (Experimental): Dexmedetomidine diluted to 10 µg/ml in Sodium Chloride 0,9 % Continuous IV infusion begun one hour before NIV session at 0.7 µg/kg/h (= 0.07 ml/kg/h) Adaptation to sedation status by changing infusion speed of 0.2 µg/kg/h (= 0.02 ml/kg/h) every 30 minutes up to 1.4 µg/kg/h (= 0.14 ml/kg/h) Sedation objective Richmond Agitation Sedation Scale -3 (moderate sedation) to 0 (alert and calm)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: DEX
Drug: Placebo
  Arms: Placebo

SUMMARY:
Crossover randomized controlled double blinded trial :

* The primary endpoint is the duration of Non Invasive Ventilation (NIV) session (minutes) with dexmedetomidine (DEX) or placebo.
* Secondary endpoints will be the sedation level as assessed by the Richmond Agitation Sedation Scale (RASS), the number of interventions to allow the completion of NIV session, the pain intensity level as assessed by visual analogue scale, the morphine and ketamine consumption during NIV sessions, the comparison of blood gas measurements before and after NIV sessions, the reproducibility of NIV cycles. The side effects of DEX will be notified.

ELIGIBILITY:
Inclusion Criteria:

* Blunt chest trauma with thoracic trauma score> 6, ICU admission and spontaneous breathing

Exclusion Criteria:

* Contra indication for NIV or Dexmedetomidine as specified by the French marketing authorization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Duration of NIV session | During ICU stay (expected average of 2 weeks)
  Minutes

SECONDARY OUTCOMES:
Richmond Agitation-Sedation Scale | During ICU stay (expected average of 2 weeks)
  From -5 (Unarousable) to +4 (Combative)
Number of interventions on NIV settings | During ICU stay (expected average of 2 weeks)
Morphine consumption | During ICU stay (expected average of 2 weeks)
  Morphine administration during NIV session (mg/kg/h)
Ketamine consumption | During ICU stay (expected average of 2 weeks)
  Ketamine administration during NIV session (mg/kg/h)
Pain visual analogue scale | During ICU stay (expected average of 2 weeks)
  From 0 (no pain) to 10 (worst pain possible)
Variation of arterial partial pressure of Carbon dioxide (CO2) before and after NIV session | During ICU stay (expected average of 2 weeks)
  mmHg
Variation of arterial partial pressure of dioxygen (O2) before and after NIV session | During ICU stay (expected average of 2 weeks)
  mmHg
Variation of potential hydrogen (pH) before and after NIV session | During ICU stay (expected average of 2 weeks)
Reproductibility of NIV sessions | During ICU stay (expected average of 2 weeks)
  Minutes
Bradycardia | During ICU stay (expected average of 2 weeks)
  Mean arterial pressure less than 55 mmHg
Hypotension | During ICU stay (expected average of 2 weeks)
  Heart rate less than 40 / mn

CONTACTS AND LOCATIONS:
Overall Officials: Thibaut TROUVE-BUISSON, PH, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU de Grenoble, Grenoble, France